CLINICAL TRIAL: NCT03422861
Title: Nabilone Use for Acute Pain in Inflammatory Bowel Disease Patients With Chronic Opioid Use Undergoing Gastrointestinal Surgery: A Single-centered Randomized Controlled Trial
Brief Title: Nabilone Use For Acute Pain in Inflammatory Bowel Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Naveed Siddiqui, Associate Professor, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NAB-2017
Record Dates: First submitted 2018-01-15; First posted 2018-02-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Nabilone; Inflammatory Bowel Disease; Opioid
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nabilone Treatment (Active Comparator): Patients who are chronic opioid users for chronic pain and have been exposed to cannabis or cannabinoid products, treated with IV PCA and nabilone as per protocol
  Interventions: Drug: Nabilone
- Placebo Treatment (Placebo Comparator): Patients who are chronic opioid users for chronic pain and have been exposed to cannabis or cannabinoid products, treated with IV PCA and placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Nabilone — Treatment regimen will involve nabilone capsule administration starting with 1mg BID orally first administered on POD #0. The patient will be continued on this medication for 72 hours
  Other Names: Cesamet
  Arms: Nabilone Treatment
Drug: Placebos — Treatment regimen will involve placebo capsule administration, identical in colour, shape, size, taste and smell to the nabilone capsules, starting orally first administered on POD #0. The patient will be continued on this medication for 72 hours
  Arms: Placebo Treatment

SUMMARY:
This is a clinical trial of nabilone for patients with Inflammatory Bowel Disease (IBD) who are undergoing IBD-related surgery (Any abdominal surgery lasting for more than one hour). This study would include a total of 80 patients undergoing general surgery who will have Intravenous Patient Controlled Analgesia (IVPCA) after surgery. It is the intention to randomize these patients postoperatively into 2 groups of 40 patients:

1. Patients who are chronic opioid users for chronic pain and have been exposed to cannabis or cannabinoid products, treated with IV PCA and nabilone as per protocol.
2. Patients who are chronic opioid users for chronic pain and have been exposed to cannabis or cannabinoid products, treated with IV PCA and placebo as per protocol.

The goal is two-fold. One is to demonstrate that patients will benefit from post-operative nabilone administration to achieve/maintain the opioid-sparing and pain modulation effects. Second is to demonstrate patients will benefit from the anti-inflammatory and immunomodulatory effects of nabilone to alleviate IBD symptoms and enhance recovery.

DETAILED DESCRIPTION:
Patients generally have pre-anesthetic visits 1-2 weeks prior to their scheduled operation. Patients identified by the Clinical Research Study Assistant (CRSA) based on inclusion and exclusion criteria will be approached regarding this study in the pre-anesthetic clinic. Patients will be made aware of the components of the study and the CRSA will be present to answer any questions. Patients have until the day of the surgery after admission to the hospital (generally 4 hours before the planned procedure) to decide whether they want to be enrolled in this study. In most cases patients will have approximately 1-2 weeks from being made aware of this study to come to a decision. Even patients who have been scheduled for pre-anesthetic clinic visit less than 1 week prior to surgery will still have >24 hrs to make decisions. Those admitted on the day of surgery may still be able to participate provided they have at least 4 hrs to review the study and have their questions answered by the study team. Patients will have access to a contact phone number in case they have additional questions. Baseline patient data will be collected once consent is obtained. On the day of surgery, administration of general anesthesia (GA) will be protocolized. Patients will cease their current oral opioid while on IV opioids. After the surgery, Patients will be randomly allocated into either placebo or intervention arm using a computerized random generator. Treatment regimen will involve nabilone capsule administration starting with 1mg twice a day orally first administered on post-operative day (POD) #0. The patient will be continued on this medication for 72 hours. Enrolled patients will document their pain scores and other data points as per study outcomes measured. The CRSA will follow for nabilone-related adverse effects at 24hrs, 48hrs, and 72hours post-operatively. Study subjects will also be followed up for psychotropic adverse reactions of nabilone (including hallucination, depressed mood, anxiety reactions, and euphoria) for 3 days after discontinuation of study treatment. This follow up will be made by the CRSA during the subject's stay in the hospital, or by telephone call made after discharge from the hospital. Any surgical complication will be recorded up to 30 days after the operation. The CRSA will administer study questionnaires and assist patients in their completion. The CRSA will work with the principal investigator (PI) to capture all requirements for study evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥25 years
* Be able to understand the study procedures
* Voluntarily provide written informed consent
* Be planned to undergo abdominal surgery related to IBD lasting more than an hour
* previously and safely tolerated side effects of nabilone use
* Chronic opioid users who are defined as opioid consumption of 20mg oral morphine equivalent per day for > 3 months
* Negative pregnancy test for females of child bearing potential and they should use acceptable birth controlling measures such as barriers, Intra Uterine Devices (IUDs) or Hormonal contraceptives consistently and correctly for one month post last dose of study drug
* Male participants must also agree to consent and correct use of acceptable contraception during and for 3 months post last dose of study drug and agree not to donate sperm during this time period (90 days)

Exclusion Criteria:

* Age under 25
* Are allergic or hypersensitive to cannabis or any cannabinoid-Have severe liver( Acute hepatitis or CHILD Score ≥2), kidney, heart (any acute condition, decompensated Heart failure or Metabolic equivalent of task(MET) < 4) or lung disease
* Have a personal or family history of serious psychotic disorders such as schizophrenia or psychosis
* Are pregnant, or are planning to get pregnant, or are breast feeding
* Are a man who wishes to start a family during duration of trial
* Have a history of alcohol or substance use disorders, including: hallucinogens (phencyclidine or similarly acting arylcyclohexylamines), other hallucinogens such as LSD, inhalants, sedatives, hypnotics, anxiolytics, and stimulants (including amphetamine-type substances, cocaine, and other stimulants).
* History of hypertension on medication
* Clinically significant lactose intolerant
* Nabilone treatment within the past month before surgery
* Diazepam or secobarbital use before surgery
* Hypersensitivity to Cesamet or any of its excipients
* Elderly (>65 years)
* History of emotional disorders

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Total amount of opioid consumption postoperatively | For up to 72 hours after surgery
  All the narcotic consumption will be converted to IV morphine equivalents using standard conversation factors

SECONDARY OUTCOMES:
Pain scores at rest and movement | Starting from discharge from post-anesthetic care unit (PACU), twice a day for 72 hours
  Based on visual analogue scale (VAS) scoring system (0-10), where score of 0 refers to no pain and a score of 10 refers to the worst pain imaginable
Incidence of opioid related side effects | Measured at 24, 48 and 72 hours
  Based on Opioid-Related Symptom Distress Scale
Incidence of nabilone side effects at 24, 48, 72 hours | Measured at 24, 48, 72 hours
  Including drowsiness, vertigo, blurred vision, sensation disturbance, dry mouth, ataxia, anorexia, asthenia, headache, orthostatic hypotension, seizure, syncope, confusion
Ulcerative Colitis (UC) symptom severity | Measured at baseline (pre-anesthetic clinic) and at 72 hrs
  Based on Simple Clinical Colitis Activity Index (SCCAI)
Crohn disease (CD) symptom severity | Measured at baseline (pre-anesthetic clinic) and at 72 hrs
  Based on Harvey-Bradshaw Index (HBI)
Time to first flatus | Assessed on a daily basis for occurrence of first flatus for up to 72 hrs
  The number of hours/days elapsed post-surgically when the patient has flatus
Number of loose stools | Measured on a daily basis for up to 72 hrs after surgery
  Predominantly watery/non-formed stool. Bristol stool chart type 6 and 7
Length of hospital stay | Measured in hours, starting from arrival to post-anesthetic care unit (PACU) to the time of discharge from hospital for up to 10 days
  The total number of hours the patient is admitted in the hospital

OTHER OUTCOMES:
Patients' Global Impression of Change (PGIC) | Measured at baseline and 72 hours
  The changes(if any) in Activity Limitations, Symptoms, Emotions and overall quality of life
Incidence of depression | Measured at baseline, 24, 48 and 72 hours and also for 72 hours after discontinuation of study treatment
  Based on Patient Health Questionnaire-9 (PHQ-9)
Incidence of psychotropic adverse reactions of Nabilone using a questionnaire | Measured for 72 hours after discontinuation of trial treatment
  We have included the most common psychotropic adverse effects of Nabilone in a questionnaire which consists of: depressed mood, euphoria, hallucination, anxiety, dissociation, suicidal ideation or behaviour
Incidence of suicide | For 72 hours after discontinuation of trial treatment
  Based on Columbia Suicide Severity Rating Scale (C-SSRS), a suicidal ideation rating scale which identifies behaviors indicative of an individual's intent to complete suicide. A "yes" answer at any time to any one of the questions necessitates further evaluation and making appropriate referrals.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, M.D, Principal Investigator — Mount Sinai Hospital Department of Anesthesia and Pain Management
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lal S, Prasad N, Ryan M, Tangri S, Silverberg MS, Gordon A, Steinhart H. Cannabis use amongst patients with inflammatory bowel disease. Eur J Gastroenterol Hepatol. 2011 Oct;23(10):891-6. doi: 10.1097/MEG.0b013e328349bb4c. PMID 21795981
- [Result] Di Sabatino A, Battista N, Biancheri P, Rapino C, Rovedatti L, Astarita G, Vanoli A, Dainese E, Guerci M, Piomelli D, Pender SL, MacDonald TT, Maccarrone M, Corazza GR. The endogenous cannabinoid system in the gut of patients with inflammatory bowel disease. Mucosal Immunol. 2011 Sep;4(5):574-83. doi: 10.1038/mi.2011.18. Epub 2011 Apr 6. PMID 21471961
- [Result] Singh UP, Singh NP, Singh B, Price RL, Nagarkatti M, Nagarkatti PS. Cannabinoid receptor-2 (CB2) agonist ameliorates colitis in IL-10(-/-) mice by attenuating the activation of T cells and promoting their apoptosis. Toxicol Appl Pharmacol. 2012 Jan 15;258(2):256-67. doi: 10.1016/j.taap.2011.11.005. Epub 2011 Nov 18. PMID 22119709
- [Result] Izzo AA, Sharkey KA. Cannabinoids and the gut: new developments and emerging concepts. Pharmacol Ther. 2010 Apr;126(1):21-38. doi: 10.1016/j.pharmthera.2009.12.005. Epub 2010 Feb 1. PMID 20117132
- [Result] Alhouayek M, Muccioli GG. The endocannabinoid system in inflammatory bowel diseases: from pathophysiology to therapeutic opportunity. Trends Mol Med. 2012 Oct;18(10):615-25. doi: 10.1016/j.molmed.2012.07.009. Epub 2012 Aug 21. PMID 22917662
- [Result] Naftali T, Lev LB, Yablecovitch D, Half E, Konikoff FM. Treatment of Crohn's disease with cannabis: an observational study. Isr Med Assoc J. 2011 Aug;13(8):455-8. PMID 21910367
- [Result] Lahat A, Lang A, Ben-Horin S. Impact of cannabis treatment on the quality of life, weight and clinical disease activity in inflammatory bowel disease patients: a pilot prospective study. Digestion. 2012;85(1):1-8. doi: 10.1159/000332079. Epub 2011 Nov 17. PMID 22095142
- [Result] Naftali T, Bar-Lev Schleider L, Dotan I, Lansky EP, Sklerovsky Benjaminov F, Konikoff FM. Cannabis induces a clinical response in patients with Crohn's disease: a prospective placebo-controlled study. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1276-1280.e1. doi: 10.1016/j.cgh.2013.04.034. Epub 2013 May 4. PMID 23648372
- [Result] Kelly S, Jhaveri MD, Sagar DR, Kendall DA, Chapman V. Activation of peripheral cannabinoid CB1 receptors inhibits mechanically evoked responses of spinal neurons in noninflamed rats and rats with hindpaw inflammation. Eur J Neurosci. 2003 Oct;18(8):2239-43. doi: 10.1046/j.1460-9568.2003.02957.x. PMID 14622184
- [Result] Ibrahim MM, Rude ML, Stagg NJ, Mata HP, Lai J, Vanderah TW, Porreca F, Buckley NE, Makriyannis A, Malan TP Jr. CB2 cannabinoid receptor mediation of antinociception. Pain. 2006 May;122(1-2):36-42. doi: 10.1016/j.pain.2005.12.018. Epub 2006 Mar 23. PMID 16563625
- [Result] Whiting PF, Wolff RF, Deshpande S, Di Nisio M, Duffy S, Hernandez AV, Keurentjes JC, Lang S, Misso K, Ryder S, Schmidlkofer S, Westwood M, Kleijnen J. Cannabinoids for Medical Use: A Systematic Review and Meta-analysis. JAMA. 2015 Jun 23-30;313(24):2456-73. doi: 10.1001/jama.2015.6358. PMID 26103030
- [Result] Salio C, Fischer J, Franzoni MF, Mackie K, Kaneko T, Conrath M. CB1-cannabinoid and mu-opioid receptor co-localization on postsynaptic target in the rat dorsal horn. Neuroreport. 2001 Dec 4;12(17):3689-92. doi: 10.1097/00001756-200112040-00017. PMID 11726775
- [Result] Smith PA, Selley DE, Sim-Selley LJ, Welch SP. Low dose combination of morphine and delta9-tetrahydrocannabinol circumvents antinociceptive tolerance and apparent desensitization of receptors. Eur J Pharmacol. 2007 Oct 1;571(2-3):129-37. doi: 10.1016/j.ejphar.2007.06.001. Epub 2007 Jun 12. PMID 17603035
- [Result] Abrams DI, Couey P, Shade SB, Kelly ME, Benowitz NL. Cannabinoid-opioid interaction in chronic pain. Clin Pharmacol Ther. 2011 Dec;90(6):844-51. doi: 10.1038/clpt.2011.188. Epub 2011 Nov 2. PMID 22048225
- [Result] Beaulieu P. Effects of nabilone, a synthetic cannabinoid, on postoperative pain. Can J Anaesth. 2006 Aug;53(8):769-75. doi: 10.1007/BF03022793. PMID 16873343
- [Result] Buggy DJ, Toogood L, Maric S, Sharpe P, Lambert DG, Rowbotham DJ. Lack of analgesic efficacy of oral delta-9-tetrahydrocannabinol in postoperative pain. Pain. 2003 Nov;106(1-2):169-72. doi: 10.1016/s0304-3959(03)00331-2. PMID 14581124
- [Result] Holdcroft A, Maze M, Dore C, Tebbs S, Thompson S. A multicenter dose-escalation study of the analgesic and adverse effects of an oral cannabis extract (Cannador) for postoperative pain management. Anesthesiology. 2006 May;104(5):1040-6. doi: 10.1097/00000542-200605000-00021. PMID 16645457
- [Result] Jain AK, Ryan JR, McMahon FG, Smith G. Evaluation of intramuscular levonantradol and placebo in acute postoperative pain. J Clin Pharmacol. 1981 Aug-Sep;21(S1):320S-326S. doi: 10.1002/j.1552-4604.1981.tb02610.x. PMID 7028791
- [Result] Von Korff M, Saunders K, Thomas Ray G, Boudreau D, Campbell C, Merrill J, Sullivan MD, Rutter CM, Silverberg MJ, Banta-Green C, Weisner C. De facto long-term opioid therapy for noncancer pain. Clin J Pain. 2008 Jul-Aug;24(6):521-7. doi: 10.1097/AJP.0b013e318169d03b. PMID 18574361
- [Result] Toth C, Mawani S, Brady S, Chan C, Liu C, Mehina E, Garven A, Bestard J, Korngut L. An enriched-enrolment, randomized withdrawal, flexible-dose, double-blind, placebo-controlled, parallel assignment efficacy study of nabilone as adjuvant in the treatment of diabetic peripheral neuropathic pain. Pain. 2012 Oct;153(10):2073-2082. doi: 10.1016/j.pain.2012.06.024. Epub 2012 Aug 23. PMID 22921260
- [Result] Turcotte D, Doupe M, Torabi M, Gomori A, Ethans K, Esfahani F, Galloway K, Namaka M. Nabilone as an adjunctive to gabapentin for multiple sclerosis-induced neuropathic pain: a randomized controlled trial. Pain Med. 2015 Jan;16(1):149-59. doi: 10.1111/pme.12569. Epub 2014 Oct 7. PMID 25288189